CLINICAL TRIAL: NCT06756191
Title: Evaluation on Efficacy and Safety of Liposomal Amphotericin B(AmBisome® ) Combination with Isavuconazole Versus AmBisome® Alone for Treatment of Patients with Pulmonary Mucormycosis
Brief Title: Antifungal Drugs in Pulmonary Mucormycosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bin Cao (Other)
Responsible Party: Sponsor-Investigator, Bin Cao, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-413
Record Dates: First submitted 2024-12-12; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Mucormycosis
Keywords: Pulmonary Mucormycosis; Amphotericin B liposome; isavuconazole
MeSH Terms: interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single drug group (Active Comparator): Liposomal amphotericin B (AmBisome®)
  Interventions: Drug: Liposomal Amphotericin B
- Combination therapy (Experimental): Liposomal amphotericin B (AmBisome®) combination with Isavuconazole
  Interventions: Drug: Combination therapy group

INTERVENTIONS:
Drug: Combination therapy group — Liposomal amphotericin B (AmBisome®) combination with Isavuconazole
  Arms: Combination therapy
Drug: Liposomal Amphotericin B — Liposomal amphotericin B (AmBisome®) alone
  Arms: Single drug group

SUMMARY:
Pulmonary mucormycosis (PM) poses a substantial clinical challenge, particularly among immunocompromised patients. The aim of the study is to determine the effectiveness and safety of administering AmBisome at a dose of 5mg/kg/day combined with isavuconazole versus using AmBisome for the management of pulmonary mucormycosis

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18 years or older diagnosed with pulmonary mucormycosis (PM).
* Individuals with Probable or proved PM, as indicated by clinical and radiological findings.

Exclusion Criteria:

* Patients with a history of pulmonary mucormycosis (PM) who have previously been treated with amphotericin B for a duration exceeding 5 days.
* Patients who have documented allergies to azoles or amphotericin B regimens
* Patients with serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or bilirubin levels exceeding five times the upper limit of normal (ULN).
* Patients with irreversible heart or liver failure, or those experiencing massive, fatal hemoptysis.
* Patients who have experienced a myocardial infarction or cerebral infarction.
* Patients currently receiving extracorporeal membrane oxygenation (ECMO) treatment.
* Pregnant or breastfeeding individuals. 8.Patients with individual reasons that may prevent them from completing the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
4-week favourable response rate | 4 week
  The percentage of patients with favourable response by 4 week. Favourable response is defined as lesion absorption in chest CT.

SECONDARY OUTCOMES:
12-week mortality | 12 week
  Defined as the proportion of patients who died by 12 week.
24-week mortality | 24 week
  Defined as the proportion of patients who died by week 24.
Frequency of adverse events | 4 week
  Treatment-related adverse event frequency

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol